CLINICAL TRIAL: NCT02963246
Title: Effects of a Mindfulness Therapy Intervention for Individuals With Inflammatory Bowel Disease: A Randomized Controlled Trial
Brief Title: Mindfulness Therapy in Inflammatory Bowel Disease
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Jose Miguel Soria Lopez, PhD, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-4
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Bowel Disease
Keywords: mindfulness; quality of life; Bowel Disease
MeSH Terms: conditions — Intestinal Diseases | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness group (Experimental): Mindfulness intervention (12 months). Mindfulness based Cognitive Therapy is an evidence-based psychological program designed to help manage depressive and stress symptoms.
  Interventions: Behavioral: Mindfulness
- Control Group (No Intervention): Treatment-as-usual control

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness-based therapy has been used effectively to treat a variety of physical and psychological disorders, including depression, anxiety, and chronic pain. Recently, several lines of research have explored the potential for mindfulness-therapy in treating somatization disorders, including fibromyalgia, chronic fatigue syndrome, and irritable bowel syndrome. Mindfulness-based therapies (MBT) are a clinical application involving the key element of nonjudgmental acceptance of physical pain or psychological distress, thereby reducing the tendency to ruminate over and catastrophise these experiences.
  In the present study, we propose a mindfulness intervention of 12 months, with sessions either personalized or online.
  Arms: Mindfulness group

SUMMARY:
Aim: To compare the effects of a specific application of Mindfulness vs. Treatment-asusual control group in patients with bowel disease. Design: randomized controlled trial. Setting: Outpatient setting. Population: patients who attended bimonthly check up.

DETAILED DESCRIPTION:
Background: Inflammatory bowel disease (IBD) is a chronic gastrointestinal condition with a relapsing disease course. Managing the relapsing nature of the disease causes daily stress for IBD patients. Mindfulness-based Cognitive Therapy (MBCT) is an evidence-based psychological program designed to help manage depressive and stress symptoms.

Aim: To compare the effects of a specific application of Mindfulness vs. Treatment-as usual control group in patients with bowel disease.

Outcome measures: quality of life, inflammatory and stress markers. Design: randomized controlled trial. Setting: Outpatient setting. Population: patients who attended bimonthly check up.

ELIGIBILITY:
Inclusion Criteria:

* patients with bowel disease diagnostic
* patients with non active disease symptoms in the last 3 month
* patients with access to internet and basic informatic knowledge

Exclusion Criteria:

* active disease symptoms
* planned surgery
* cognitive impairment
* previous experience with mindfulness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Quality of life measured with the IBDQ-32 (Inflammatory Bowel Disease Questionnaire) | Change from Baseline IBDQ-32 score at 12 months

SECONDARY OUTCOMES:
inflammation stress markers (reactive Protein C and faecal calprotectin) | Change from Baseline inflammation stress markers at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: José M Soria, PhD, Principal Investigator — University CEU Cardenal Herrera. Plaza Reyes Católicos nº19 03204 Elche, Alicante, Spain
Locations (1):
- Universidad CEU Cardenal Herrera, Elche, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391